CLINICAL TRIAL: NCT06656741
Title: Neurological Evidence of Diverse Self-Help Breathing Trainings with Virtual Reality and Bio-Feedback Assistance: an Extensive Exploration of EEG Markers
Brief Title: Neurological Evidence of Diverse Self-Help Breathing Trainings with Virtual Reality and Bio-Feedback Assistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hei-Yin Hydra Ng (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, Hei-Yin Hydra Ng, Principal Investigator, National Tsing Hua University
Organization: National Tsing Hua University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NCTU-REC-109-037F; MOST 110-2636-E007-018 (Other Grant/Funding Number: Ministry of Science and Technology of Taiwan)
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Breath Training Styles
Keywords: bio-feedback; virtual reality; breath training; EEG; effective connectivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single group (Experimental): This is a single group study. All participants belong to this group. Participants will perform resting state task, mindful breathing task, guided breath task, and breath counting task respectively. The task sequence is counter-balanced.
  Interventions: Behavioral: Resting State; Behavioral: Mindful Breathing; Behavioral: Guided Breathing; Behavioral: Breath Counting

INTERVENTIONS:
Behavioral: Resting State — Resting state is a mental state and a research paradigm that people do nothing and idle as much as possible to show their baseline neuro signals. In this task, we instructed participants to rest with their eyes opened for 6 minutes. The VR environment of blue sky and swaying meadow was presented to the participants throughout this task.
Behavioral: Mindful Breathing — Mindful breathing is a state that people focus on their inner sensation. In this task, the meadow's motion in the VR environment corresponded to the participants' inhalation and exhalation, as detected by the respiration belt. The participants were instructed to focus mentally on their bodily sensations as they breathed, with the meadow's sway as a visual cue.
Behavioral: Guided Breathing — Guided breathing refers to the breath training technique that trainees are guided to inhale and exhale according to a fixed tempo. In this task, meadow swayed in a fixed tempo of 4 seconds back and 6 seconds forth. The participants were instructed to synchronize their inhalation with the meadow's backward motion (lasting 4 seconds) and their exhalation with its forward motion (lasting 6 seconds).
Behavioral: Breath Counting — Breath counting refers to the breath training technique that trainees mentally count the numbers of breath cycles they have finished in a certain period of time. In this task, similar to the mindful breathing task, the meadow's motion was synchronized with the participants' breathing patterns. During the 6 minutes, we instructed the participants to breathe naturally and mentally count their breathing cycles.

SUMMARY:
The goal of this research is to learn about the neuro-mechanism beneath breath training, mindfulness meditation, or periods of idleness. This research also focuses on the use of virtual reality (VR) and bio-feedback (BF) integrated assistance system in breath training, and seeks for the potential of generalizing breath training in public.

The main questions it aims to answer are:

Whether and how people's neuro-mechanism (indicated by EEG indexes) changes when they are performing different breath training techniques (i.e., mindful breathing, guided breathing, and breath counting).

Researchers will compare the neuro-markers when participants perform different styles of breath training.

Participants will:

* Participants will equip an EEG system, a VR headset, a respiratory belt, and a heartbeat sensor.
* Participants will perform resting state task, mindful breathing task, guided breath task, and breath counting task respectively.
* EEG activity, breath rate, reaction time, accuracy, and HRV will be recorded. Each session will last approximately two hours.

DETAILED DESCRIPTION:
1. Research Overview In today's fast-paced industrial society, managing individual physical and psychological stress has become crucial for maintaining mental, emotional, and brain health. Practices such as breath training, mindfulness meditation, or periods of idleness have been suggested as effective means to relieve stress, reduce anxiety, and improve sleep quality. This study combines cognitive psychology behavioral measurements, electroencephalography (EEG), and heart rate variability (HRV) to investigate the cognitive function, brain structure, and brain activity of adults with breath training/mindfulness meditation experience or regular episodes of mind-wandering. Meanwhile, this research also focuses on the use of technology, namely virtual reality (VR) and bio-feedback (BF) integrated assistance system, and seeks for the potential of generalizing breath training in public. By utilizing non-invasive neuroimaging techniques, this research aims to provide scientific evidence regarding the effects of breath training/mindfulness meditation and mind-wandering. Ultimately, the study seeks to apply these findings to improve national mental and brain health.

   The research questions are: whether and how people's neuro-mechanism (indicated by EEG indexes) changes when they are performing different breath training techniques (i.e., mindful breathing, guided breathing, and breath counting).
2. Research Participants Age range: 20-80 years old. Total: 53 participants.

   Withdrawal Criteria:

   Participants can withdraw at any point if they feel discomfort.
3. Compensation for Participation: Participants will receive a total of NT$1,000.
4. Informed Consent Process The research personnel will explain the study to participants at the study locations. The informed consent process will take approximately 30 minutes per participant.
5. Potential Side Effects, Follow-Up Procedures, and Necessary Rehabilitation Plans

   1. Physiological Risks:

      • Electroencephalography (EEG): EEG measures brain activity passively from the scalp using a non-invasive method that does not involve electrical discharge or radiation, thus posing no harm to participants. During the application of conductive gel with blunt needles, the needles may touch the scalp but will not cause any damage. All needles are sterilized with alcohol before use. Participants are encouraged to notify the experimenter immediately if any discomfort arises. The gel will remain on the participant's scalp throughout the experiment, and electrodes around the eyes will be affixed using breathable medical tape. For individuals with sensitive skin, mild itching may occur, although no allergic reactions have been reported.
   2. Psychological Risks:

      There is a minimal risk of psychological discomfort during the study. Participants may discontinue the experiment at any time if they feel uncomfortable.
   3. Social Risks:

   Participants may face minimal social risks, but the research team will make every effort to protect their privacy and confidentiality in accordance with legal requirements.
6. Privacy and Data Confidentiality

   1. All collected data and samples will be securely locked, and electronic data will be stored on password-protected systems.
   2. Data Preservation and Confidentiality:

      * Participant data, including names and other identifiable information, will be coded or anonymized (e.g., using initials).
      * The "de-identification" method will ensure that no linkages to identifiable information can be made in the future.
   3. Handling of Remaining Samples and Confidential Data After Study Completion:

      * Identifiable data will be destroyed by the principal investigator five years after the study ends (December 31, 2028).
      * EEG data will be anonymized and preserved for future research, with all identifiable links permanently removed. No identifying information will appear in any published academic articles.
7. Research Procedures This cross-sectional study will use various cognitive psychology paradigms and EEG to examine cognitive function, brain activity, and structure in adults. Participants will complete self-report questionnaires regarding their mental and physiological states.

   Participants will equip an EEG system, a VR headset, a respiratory belt, and a heartbeat sensor. Participants will perform resting state task, mindful breathing task, guided breath task, and breath counting task respectively, with the sequence counter-balanced. EEG activity, breath rate, reaction time, accuracy, and HRV will be recorded. Each session will last approximately two hours.
8. Evaluation and Statistical Methods EEG data will be analyzed using MATLAB and SPM (Statistical Parametric Mapping), with statistical analyses performed in SPSS. Brain activation and structural data will be evaluated, and ANOVA will be applied to questionnaires and behavioral data. Relationships between behavioral and neural measures will be examined, and statistical significance will be determined at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged between 20 and 80.
2. Normal vision or corrected-to-normal vision.

Exclusion Criteria:

1. History of epilepsy, brain injury, or other neurological disorders in the individual or their family.
2. Long-term use of medication (e.g., antidepressants, sleep aids).
3. Claustrophobia.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
EEG effective connectivity(dDTF) | Through study completion, an average of 1 hour
  This study employed the direct directed transfer function (dDTF) to evaluate causal relationships between EEG channels. Modified from the directed transfer function, the dDTF is an effective connectivity estimator grounded in frequency-domain Granger causality. The dDTF isolates and assesses the direct causal link between a specific pair of channels, effectively mitigating the impact of indirect neural influences because of brain tissue conductivity.
EEG connectivity inflow | Through study completion, an average of 1 hour
  For a given EEG channel, the connectivity inflow represents the cumulative sum of all corresponding incoming connectivity edges.
EEG connectivity outflow | Through study completion, an average of 1 hour
  For a given EEG channel, the connectivity outflow represents the cumulative sum of all corresponding outgoing connectivity edges.
EEG band power | Through study completion, an average of 1 hour
  We converted the EEG data to a frequency-domain signal using a short-time Fourier transformation. All transformed spectra were then log-transformed and represented in dB (10log10).

OTHER OUTCOMES:
EEG activity | Through study completion, an average of 1 hour
  A Brain Products GmbH 32-channel LiveAmp EEG system (Gilching, Germany) was used to collect the EEG data at a sampling rate of 1,000 Hz and a resolution of 40.7 nV. We mounted the electrodes on a Brain Products EasyCap (Gilching, Germany), the layout of which followed the international 10/20 electrode placement system. The electrode-skin impedance was maintained under 10 kΩ with an abrasive electrode paste (Abralyt HiCl). EEG data on all channels were acquired using FCz as the reference and were filtered using a band-pass filter of 0.0159 Hz and 250 Hz, plus a 60 Hz notch filter.
Breath rate | Through study completion, an average of 1 hour
  A Vernier Go Direct® Respiration Belt (Beaverton, Oregon, U.S.) monitored and captured the respiration data at a sampling rate of 1,000 Hz. The respiration belt was worn on the rib cage. After the initiation of each experimental condition (i.e., each breathing technique), the program collected 10 seconds of a respiratory signal from each participant for normalization. We compared the respiratory signal with the normalized signal to determine whether the participant was inhaling or exhaling.
Heart rate | Through study completion, an average of 1 hour
  The ArtiseBio Cygnus-819997-RawEEG system (Hsinchu, Taiwan) was employed to collect ECG data at a sampling rate of 1,000 Hz. Three electrodes from the ArtiseBio system were affixed to Kendall 200 series electrode pads (Cardinal Health, Dublin, Ohio, U.S.) and positioned according to the standard limb leads II configuration for heart rate monitoring.
Five Facet Mindfulness Questionnaire | 1 day
  Five Facet Mindfulness Questionnaire (FFMQ) is measure of people's mindfulness level. FFMQ consists of 39 items, and the score ranges between 1 and 39. The higher score represents the higher mindfulness level.
Montreal Cognitive Assessment | 1 day
  Montreal Cognitive Assessment (MoCA) is a questionnaire for the early detection of mild cognitive impairment. MoCA consists of 30 items, and the score ranges between 0 and 30. The higher score represents the better cognitive function.
Beck Depression Inventory | 1 day
  Beck Depression Inventory (BDI) is a self-report measure of people's symptoms of depression. BDI consists of 21 items, and the score ranges between 0 to 21. The higher score represents the higher depression level.
Beck Anxiety Inventory | 1 day
  Beck Anxiety Inventory (BAI) is a self-report measure of people's symptoms of anxiety. BAI consists of 21 items, the score ranges between 0 to 21. The higher score represents the higher anxiety level.
Mind Wandering Questionnaire | 1 day
  Mind Wandering Questionnaire measures people's frequency of mind-wandering. It consists of 5 items, the score ranges between 1 and 30. The higher score represents more frequent mind-wandering.
Pittsburgh Sleep Quality Index | 1 day
  Pittsburgh Sleep Quality Index (PSQI) is a self-report measurement of people's sleep difficulty. It consists of 9 items, the score ranges between 1 and 21. The higher score represents the higher level of sleep difficulty.

CONTACTS AND LOCATIONS:
Locations (1):
- National Tsing Hua University, Hsinchu, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No
National Yang Ming Chiao Tung University - Research Ethics Center for Human Subject Protection (NYCU-REC) reviewed and approved this study (Project Number: NCTU-REC-109-037F). In accordance with the regulations of NYCU-REC, only the project-related personnel, as listed in NYCU-REC (Project Number: NCTU-REC-109-037F), may access the individual participant data.

REFERENCES:
- [Background] Lukic YX, Teepe GW, Fleisch E, Kowatsch T. Breathing as an Input Modality in a Gameful Breathing Training App (Breeze 2): Development and Evaluation Study. JMIR Serious Games. 2022 Aug 16;10(3):e39186. doi: 10.2196/39186. PMID 35972793
- [Background] Luddecke R, Felnhofer A. Virtual Reality Biofeedback in Health: A Scoping Review. Appl Psychophysiol Biofeedback. 2022 Mar;47(1):1-15. doi: 10.1007/s10484-021-09529-9. Epub 2021 Dec 3. PMID 34860290
- [Background] Giggins OM, Persson UM, Caulfield B. Biofeedback in rehabilitation. J Neuroeng Rehabil. 2013 Jun 18;10:60. doi: 10.1186/1743-0003-10-60. PMID 23777436
- [Derived] Ng HH, Wu CW, Hsu HC, Huang CM, Hsu AL, Chao YP, Jung TP, Chuang CH. Neurological Evidence of Diverse Self-Help Breathing Training With Virtual Reality and Biofeedback Assistance: Extensive Exploration Study of Electroencephalography Markers. JMIR Form Res. 2024 Dec 6;8:e55478. doi: 10.2196/55478. PMID 39642375